CLINICAL TRIAL: NCT06253078
Title: Ciprofol EC50 for Inducing Loss of Consciousness in Elderly Patients: an Exploratory Study Based on Dixon's Up-and-Down Method
Brief Title: Ciprofol EC50 for Inducing Loss of Consciousness in Elderly Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2024-76（IIT）
Record Dates: First submitted 2024-01-29; First posted 2024-02-12 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Elderly Patients
Keywords: Ciprofol; EC50; Los of consciousness; Elderly; General anesthesia
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 65-69 years old (Experimental): The initial dose of ciprofol was 0.4mg/ in this group.
  Interventions: Drug: Ciprofol dose 0.4mg/Kg
- 70-74 years old (Experimental): The initial dose of ciprofol was 0.4mg/ in this group.
  Interventions: Drug: Ciprofol dose 0.4mg/Kg
- 75-79 years old (Experimental): The initial dose of ciprofol was 0.3mg/ in this group.
  Interventions: Drug: Ciprofol dose 0.3mg/Kg
- 80-84 years old (Experimental): The initial dose of ciprofol was 0.3mg/ in this group.
  Interventions: Drug: Ciprofol dose 0.3mg/Kg
- Older than 85 years (include 85 years old) (Experimental): The initial dose of ciprofol was 0.2mg/ in this group.
  Interventions: Drug: Ciprofol dose 0.2mg/Kg

INTERVENTIONS:
Drug: Ciprofol dose 0.4mg/Kg — The initial dose of ciprofol was 0.4mg/Kg for induction in this group.
  Other Names: 0.4mg/Kg ciprofol
  Arms: 65-69 years old; 70-74 years old
Drug: Ciprofol dose 0.3mg/Kg — The initial dose of ciprofol was 0.3mg/Kg for induction in this group.
  Other Names: 0.3mg/Kg ciprofol
  Arms: 75-79 years old; 80-84 years old
Drug: Ciprofol dose 0.2mg/Kg — The initial dose of ciprofol was 0.2mg/Kg for induction in this group.
  Other Names: 0.2mg/Kg ciprofol
  Arms: Older than 85 years (include 85 years old)

SUMMARY:
ciprofol is a recently introduced novel sedative drug. In comparison to the traditional propofol, ciprofol exhibits a higher affinity for GABA A receptors, approximately 4-5 times that of propofol, and possesses fewer side effects, particularly notable in respiratory depression and injection pain. In the context of general anesthesia induction, recent research has confirmed a 100% success rate in the induction of general anesthesia for elderly patients (65-80 years old) undergoing non-cardiac surgery with a dosage range of 0.2mg/kg-0.4mg/kg ciprofol. However, for elderly patients aged 65 and above, even up to 85 years old, it is currently not entirely clear what dosage should be selected for patients in different age groups. Consequently, we have designed this trial with the aim of exploring the dosage requirements of ciprofol during general anesthesia induction among elderly patients in various age brackets.

Methods: This is a prospective, non-controlled, non-randomized, single-blind study. Elderly patients aged 65 years and older were enrolled in the study with American Society of Anesthesiologists (ASA) physical status I or II undergoing general anesthesia. All patients were divided into five groups according to age, and the corresponding initial dose of ciprofol administered was selected according to the grouping, with subsequent doses of ciprofol determined according to the Dixon up-and-down method. At least seven crossover points were obtained before the conclusion of the study.The primary outcomes were the dose of ciprofol administered at the time of loss of consciousness (mg/Kg) and the plasma concentration of ciprofol.

DETAILED DESCRIPTION:
After received the approvement of ethics committee of the Cancer Hospital of the University of Chinese Academy of Sciences (approval number IRB-2024-76(IIT)). The study was registered before patient enrollment in Clinicaltrials.Written informed consent was obtained from all participants. The study was performed from Jan 1, 2024 to Dec 31, 2025. 150 patients aged 65 years and above, ASA physical status I or II, undergoing surgery under general anesthesia and who were not allergic to the study drug were included in this study. Basic monitoring such as 3-lead electrocardiogram, pulse oximetry, and noninvasive blood pressure were arranged preoperatively. All patients were divided into five groups according to age, The initial dose of ciprofol for the first elderly patient was 0.2-0.4 mg/kg, the initial concentration was 0.4 mg/Kg for patients aged 65-74 years, 0.3 mg/Kg for patients aged 75-84 years, and 0.2 mg/Kg for patients aged 85 years or older, and the ciprofol doses for adjacent patients were set to be equidistantly spaced up and down by 0.05 mg/kg. Evaluation of the eyelash reflex and speech reflex was performed after intravenous infusion of ciprofol to observe whether LOC occurred within 4 min. After loss of consciousness, sufentanil (5ug/ml, diluted in 0.9% saline) and rocuronium bromide were given for endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* 65 ≤ age years;
* ASA physical state I and II;
* Hadn't a history of allergy to the drugs used in this study;

Exclusion Criteria:

* America Society of Anesthesiologists (ASA) class >III;
* Allergic to anesthetic solutions or the drugs used in this study;
* Body mass index (BMI) ≤ 20 or ≥ 30 kg/m2;
* Using hypnotics, opioid analgesics, or anti-anxiety medications;
* Known or suspected heart failure (ejection fraction <40%), severe respiratory disease, renal or metabolic disease
* Refuse to participate or participate with other clinical investigators ;

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ciprofol EC50 (mg/Kg) for loss of consciousness | From loss of consciousness (LOC) to 10 minutes after trachea intubation.
  Use up-and-down method to evaluate the Ciprofol EC50 for loss of consciousness in different age groups.

SECONDARY OUTCOMES:
Plasma concentration of ciprofol when LOC. | From the start of induction to loss of consciousness, approximately 4 to 8 minutes after start of induction.
  Measure the plasma concentration of ciprofol when LOC.
The mean artery pressure | From entering the OR to 10 minutes after trachea intubation.
  Hemodynamic fluctuation during induction
The heart rate | From entering the OR to 10 minutes after trachea intubation.
  Hemodynamic fluctuation during induction
Incidence of adverse events | From entering the OR to 10 minutes after trachea intubation.
  Measuring and recording the adverse events such as hypotension, hypertension, bradycardia and tachycardia during induction period.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, Dr., Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Jiangling Wang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Plan can be shared when required.